CLINICAL TRIAL: NCT03050593
Title: Prospective, Observational, Single-centre, Cohort Study Aimed at Developing Imaging and Plasma Biomarkers in Heart Failure With Preserved Ejection Fraction
Brief Title: Developing Imaging And plasMa biOmarkers iN Describing Heart Failure With Preserved Ejection Fraction (DIAMONDHFpEF)
Acronym: DIAMONDHFpEF
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0328
Record Dates: First submitted 2017-02-06; First posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2015-05

CONDITIONS: Patients With Heart Failure and Preserved Ejection Fraction - HFpEF; Patients With Heart Failure With Reduced Ejection Fraction - HFrEF; Healthy Controls Group - Age and Sex-matched
Keywords: HFpEF; HFrEF
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA Plasma, serum, urine, DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HFpEF group: clinical or radiographic evidence of heart failure and left ventricular ejection fraction > 50% on transthoracic echocardiography
  Interventions: Diagnostic Test: MRI scan, Echo scan
- HFrEF group: Clinical or radiographic evidence of heart failure and left ventricular ejection fraction < 40% on transthoracic echocardiography
  Interventions: Diagnostic Test: MRI scan, Echo scan
- Healthy control group: Asymptomatic controls (age and sex-matched) without known heart disease
  Interventions: Diagnostic Test: MRI scan, Echo scan

INTERVENTIONS:
Diagnostic Test: MRI scan, Echo scan
  Other Names: cardiac MRI, trans thoracic echocardiography

SUMMARY:
The investigators wish to test a hypothesis that patients with HFpEF have different characteristics on echo, cardiac MRI and plasma protein & chemical profiles compared to HFrEF and healthy volunteers.

DETAILED DESCRIPTION:
Large scale prospective studies incorporating cardiac MRI, echocardiography and plasma sampling are currently lacking in HFpEF. The main aims of our study are to:

1. better phenotype and characterise HFpEF (also comparing with HFrEF and age- and sex- matched healthy controls)
2. provide mechanistic insights into pathophysiology
3. describe potential biomarkers and their relation to relevant clinical outcomes (exercise capacity, heart failure quality of life and prognosis)

ELIGIBILITY:
Inclusion Criteria:

* Clinical features of heart failure or prior radiographic evidence in the absence of symptoms And Either ejection fraction > 50% (for HFpEF arm) or ejection fraction < 40% (for HFrEF arm)

Exclusion Criteria:

* Myocardial infarction within the preceding 6 months
* Suspected or confirmed cardiomyopathy (e.g. hypertrophic, infiltrative)
* Suspected or confirmed constrictive pericarditis
* Significant native valve disease (≥ moderate severity)
* Known Significant lung disease (documented or FEV1< 30% or FVC < 50%)
* Non-cardiovascular co-morbidity likely to cause death within 6 months (e.g. malignancy)
* Significant renal failure (estimated GFR < 30 ml/min/m2)
* Patient inability to provide informed consent (e.g. dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with heart failure from Hospital (including ward patients and out-patients clinic)
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The composite end-point of all-cause mortality or repeat hospitalisation with heart failure | Minimum 6 month follow-up

SECONDARY OUTCOMES:
The number of new clinical diagnoses detected by cardiac MRI | Through study completion, an average of 1 year
Exercise capacity as assessed by the six-minute walk test | Through study completion, an average of 1 year
Quality of life assessed by the Minnesota Living with Heart Failure Questionnaire | Through study completion, an average of 1 year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arnold JR, Kanagala P, Budgeon CA, Jerosch-Herold M, Gulsin GS, Singh A, Khan JN, Chan DCS, Squire IB, Ng LL, McCann GP. Prevalence and Prognostic Significance of Microvascular Dysfunction in Heart Failure With Preserved Ejection Fraction. JACC Cardiovasc Imaging. 2022 Jun;15(6):1001-1011. doi: 10.1016/j.jcmg.2021.11.022. Epub 2022 Jan 12. PMID 35033490
- [Derived] Kanagala P, Arnold JR, Khan JN, Singh A, Gulsin GS, Chan DCS, Cheng ASH, Yang J, Li Z, Gupta P, Squire IB, McCann GP, Ng LL. Plasma Tenascin-C: a prognostic biomarker in heart failure with preserved ejection fraction. Biomarkers. 2020 Nov;25(7):556-565. doi: 10.1080/1354750X.2020.1810319. Epub 2020 Aug 28. PMID 32803990
- [Derived] Kanagala P, Arnold JR, Singh A, Khan JN, Gulsin GS, Gupta P, Squire IB, Ng LL, McCann GP. Prevalence of right ventricular dysfunction and prognostic significance in heart failure with preserved ejection fraction. Int J Cardiovasc Imaging. 2021 Jan;37(1):255-266. doi: 10.1007/s10554-020-01953-y. Epub 2020 Jul 31. PMID 32737707
- [Derived] Gulsin GS, Kanagala P, Chan DCS, Cheng ASH, Athithan L, Graham-Brown MPM, Singh A, Yang J, Li Z, Khunti K, Davies MJ, Arnold JR, Squire IB, Ng LL, McCann GP. Differential left ventricular and left atrial remodelling in heart failure with preserved ejection fraction patients with and without diabetes. Ther Adv Endocrinol Metab. 2019 Jul 5;10:2042018819861593. doi: 10.1177/2042018819861593. eCollection 2019. PMID 31308926
- [Derived] Kanagala P, Cheng ASH, Singh A, Khan JN, Gulsin GS, Patel P, Gupta P, Arnold JR, Squire IB, Ng LL, McCann GP. Relationship Between Focal and Diffuse Fibrosis Assessed by CMR and Clinical Outcomes in Heart Failure With Preserved Ejection Fraction. JACC Cardiovasc Imaging. 2019 Nov;12(11 Pt 2):2291-2301. doi: 10.1016/j.jcmg.2018.11.031. Epub 2019 Feb 13. PMID 30772227
- [Derived] Kanagala P, Cheng ASH, Singh A, McAdam J, Marsh AM, Arnold JR, Squire IB, Ng LL, McCann GP. Diagnostic and prognostic utility of cardiovascular magnetic resonance imaging in heart failure with preserved ejection fraction - implications for clinical trials. J Cardiovasc Magn Reson. 2018 Jan 11;20(1):4. doi: 10.1186/s12968-017-0424-9. PMID 29321034